CLINICAL TRIAL: NCT04205994
Title: Dopaminergic Mechanisms Underlying Human Social Behavior: A Multimodal Approach
Brief Title: Dopaminergic Mechanisms Underlying Human Social Behavior
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: University of California, San Francisco (Other); Lawrence Berkeley National Laboratory (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 231378
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Decision Making; Executive Function; Dopamine
MeSH Terms: interventions — Tolcapone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tolcapone (Experimental): Tolcapone is a brain penetrant catechol-O-methyltransferase (COMT) inhibitor. It will be administered in a single 200mg dosage once in randomized, double-blind, counterbalanced fashion with a placebo.
  Interventions: Drug: Tolcapone 200 MG; Other: Functional Magnetic Resonance Imaging (fMRI)
- Placebo (Placebo Comparator): Placebo will be administered in a single pill once in randomized, double-blind, counterbalanced fashion with a placebo.
  Interventions: Other: Functional Magnetic Resonance Imaging (fMRI)

INTERVENTIONS:
Drug: Tolcapone 200 MG — Tolcapone is a brain penetrant catechol-O-methyltransferase (COMT) inhibitor. It will be administered in randomized, double-blind, counterbalanced fashion with a placebo.
  Arms: Tolcapone
Other: Functional Magnetic Resonance Imaging (fMRI) — FMRI provides an indirect and noninvasive measure of brain activity.

SUMMARY:
Developing theoretical, quantitative models of the basic cognitive mechanisms underlying human social decision-making, and understanding the influence of neuromodulators such as dopamine on these mechanisms, has important ramifications for both healthy and patient populations. In this proposal the investigators combine quantitative social measures, computational models, neuroimaging, and a pharmacological intervention to define the mechanisms of social decision-making.

DETAILED DESCRIPTION:
A significant challenge for understanding social dysfunctions observed in mental illness is to link high-level theories of social behavior and cognition with the computations performed by brain circuits. Specifically, how does the brain translate social perception into social valuation, and how does such valuation influence social actions? Investigators propose to leverage recent developments in economic theory and cognitive neuroscience to bridge this divide using a computational, model-based approach. In this proposal, investigators hypothesize that social behavior is underpinned by brain mechanisms that are influenced by the neurotransmitter dopamine, and that these mechanisms can be captured by computational models that integrate internal representations of social experience, and parameters relevant to dopamine tone, to inform social actions. Social valuation thus critically, and quantitatively, depends upon both internal social representations and the neurochemistry of the actor within the social environment. To assess this hypothesis, investigators pursue two approaches to evaluate dopamine tone: one in which investigators use an FDA-approved medication, tolcapone, to influence dopamine metabolism, and one in which investigators perform Positron Emission Tomography (PET) imaging to measure dopamine release and baseline dopamine receptor D2/D3 occupancy. Investigators then apply a model of social valuation to subjects' behavior, and search for neural correlates of this valuation using functional MRI (fMRI). To this end, investigators bring together a group of experts in (1) the neuroeconomics and modeling of social and non-social decision-making, (2) cognitive neuroscience, (3) the pharmacology of frontostriatal circuits, and (4) neuroimaging. Investigators thus seek to broaden our understanding of the computations and circuits underlying social behavior. Moreover, investigators believe that a model-based understanding of these behaviors and neural circuits may guide more robust predictions of the effects of pharmacological manipulations on social valuation, and provide quantitative tools to assess the effects of such manipulations in patient populations, with possible therapeutic implications.

ELIGIBILITY:
Inclusion criteria:

* Ages 18-40 and right-handed
* Able to provide written informed consent
* Normal or corrected-to-normal visual acuity
* General good health as determined for tolcapone studies by screening provider (Dr. Kayser, Dr.Jagust, or other approved, licensed clinician)

Exclusion criteria:

* Regular and/or scheduled use of other neuro- or psycho-active medications
* Severe low blood pressure or uncontrolled high blood pressure
* Intelligence quotient (IQ) < 70 as assessed by the Wechsler Test of Adult Reading (WTAR)
* History of mild, moderate, or severe traumatic brain injury
* History of brain surgery (i.e. violating brain parenchyma) or penetrating brain injury
* Active alcohol dependence or alcohol abuse by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria (within previous 30 days)
* Active substance dependence or substance abuse by DSM-IV-TR criteria (excluding nicotine, but including marijuana, opiates, stimulants (cocaine, amphetamines), and hallucinogens within previous 30 days)
* History of suicide attempt (last 5 years)
* Clinically severe medical illness requiring treatment
* History of brain tumor, stroke, demyelinating disease, encephalitis, or cerebral aneurysm rupture
* Clinical diagnosis of Alzheimer's disease or other primary neurodegenerative disorder
* Schizophrenia or other psychiatric disturbances

For Subjects Undergoing fMRI Scanning:

* Contraindications to MRI (e.g. unremovable ferromagnetic metals, claustrophobia)
* Inability to complete basic fMRI requirements (e.g. to make button presses and to minimize movement < 5mm)
* Women of childbearing potential take a urine pregnancy test prior to scanning.

For Tolcapone Experiments:

* Contraindications to tolcapone use, including liver function tests elevated more than 2.5 times above normal ranges, pregnancy, previous adverse reaction to tolcapone, significant liver or kidney impairment
* Current use (within previous 30 days) of pharmacological agents with dopaminergic actions, including but not limited to levodopa/carbidopa, entacapone, tolcapone, amantadine, bromocriptine, pergolide, pramipexole, ropinirole, selegiline, isocarboxazid, phenelzine, tranylcypromine, clozapine, olanzapine, quetiapine, risperidone, ziprasidone, aripiprazole, fluphenazine, haloperidol, perphenazine, pimozide, thiothixene, trifluoperazine, loxapine, molindone, chlorpromazine, mesoridazine, thioridazine, promethazine, dextroamphetamine, dexmethylphenidate, dextroamphetamine, or methylphenidate

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Behavioral responses in neuroeconomic tasks | Up to 4 weeks
  Subjects will make financial decisions involving themselves and another person in the context of model-based neuroeconomic games.
Blood oxygen level dependent (BOLD) activity | Up to 4 weeks
  BOLD activity represents an indirect measure of brain activity, and will be correlated with behavioral task performance.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hsu, PhD, Principal Investigator — University of California, Berkeley
Locations (1):
- University of California, Berkeley, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data and software code will be posted and shared via Open Science Foundation.
Supporting Information: Analytic Code
Time Frame: We anticipate posting the data and code 2 years following completion of study on Open Science Foundation. All data and code will be anonymized to ensure confidentiality of participants. The data and code will be available indefinitely once posted.
Access Criteria: Data and code will be public access once posted.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/94/NCT04205994/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/94/NCT04205994/ICF_001.pdf